CLINICAL TRIAL: NCT05134363
Title: Dexmedetomidine for Prophylaxis Against Postoperative Nausea and Vomiting in Highly Susceptible Patients: a Randomised Controlled Comparison of Two Bolus Doses
Brief Title: Dexmedetomidine for Prophylaxis Against PONV in Highly Susceptible Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Raafat Mahmoud Seif, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD-208-2021
Record Dates: First submitted 2021-10-30; First posted 2021-11-24 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Nausea and Vomiting; Head and Neck Surgeries
Keywords: Dexmedetomidine; PONV; ondansetron; post operative; nausea; vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: comparative study between two doses and a 3rd control group
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine 0.5 mic/kg bolus (Active Comparator): selective alpha 2 adrenergic receptor agonist
  Interventions: Drug: Dexmedetomidine Hydrochloride 0.5 mic/kg bolus
- dexmedetomidine 0.75 mic/kg bllus (Active Comparator): selective alpha 2 adrenergic receptor agonist
  Interventions: Drug: Dexmedetomidine Hydrochloride 0.75 mic/kg bolus
- Placebo group (Placebo Comparator): receving equal volume of normal saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride 0.5 mic/kg bolus — comparison between two bolus doses of dexmedetomidine with a placebo group
  Arms: Dexmedetomidine 0.5 mic/kg bolus
Drug: Dexmedetomidine Hydrochloride 0.75 mic/kg bolus — comparison between two bolus doses of dexmedetomidine with a conventional group receiving ondansetron.
  Arms: dexmedetomidine 0.75 mic/kg bllus
Drug: Placebo — equal volume of normal saline
  Arms: Placebo group

SUMMARY:
The study aims to compare between two bolus doses of dexmedetomidine in preventing PONV in highly susceptible patients.

DETAILED DESCRIPTION:
Being A challenging complaint, many studies tried to find an effective preventive strategies for PONV. In this study protocol the investigators aim to compare between 0.5 mic/kg and 0.75 mic/kg bolus doses of dexmedetomidine when given toward the end of head and neck surgeries in highly susceptible patients with a controlled group receiving ondansetron.

The primary outcome is the 1st 24 hours incidence of PONV

Other outcomes include:

* Time to 1st call for rescue antiemetic and the total amount of antiemetics
* Number of PONV attacks
* Post operative pain score with visual analogous scale (VAS) and time to 1st call for rescue analgesia
* Sedation Score using Observer's Assessment of Alertness and sedation (OAA/S)
* Patient satisfaction
* Vital signs in the 1st 24 hours

ELIGIBILITY:
Inclusion Criteria:

* Two risk factors or more for PONV ( female, non-smoking, postoperative opioids, history of motion sickness or PONV )
* Head and neck surgeries in adults
* ASA ( I , II )

Exclusion Criteria:

* Patients on ( steroids , antiemetics or any drug caude emesis )
* Any active cardiac condition at the time of the surgery
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV in the 1st 24 hours postoperatively | The first 24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  The overall incidence of nausea and vomiting in the 1st 24 hours following Head and neck surgeries.

SECONDARY OUTCOMES:
Number of PONV attacks | The first24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  Number of PONV attacks in the 1st 24 hours following Head and neck surgeries
Pain score postoperatively. | The first24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  Pain assessement using visual analogous scale score (0-10) with 10 denoting the worst pain expressed and zero= no pain
Sedation score | The first24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  using Observer's assessment of ALERTNESS and Sedation (1-5)with 1 = unconscious and 5= Alert
Patient satisfaction | The first24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  The patient completes a simple questionnaire with 0= very satisfied 1 = satisfied 2= not satisfied
Blood pressure | The first24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  Mean arterial blood pressure (MAP) in the 1st 24 hours
Heart Rate (HR) | The first24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  Pulse rate in the 1st 24 hours
The time to 1st call for rescue antiemetic | In the 1st 24 hours
  time to 1st call for rescue antiemetic and the severity of nausea ( using the 11 verbal 11-point rating scale 0= no nausea 10= the worst nausea
The severity of nausea. | The first24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  the severity of nausea ( using the 11 verbal 11-point rating scale 0= no nausea 10= the worst nausea
Total amount of morphine consumption | The first24 hours ( every half an hour in the 1st 2 hours and then at 4,6,8,12 and 24 hours )
  morphine consumed in thw 1st 24 hours in milligrams.
The time to 1st call for rescue analgesia | In the first 24 hours
  time to 1st call for rescure analgesic medication in the 1st 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apfel CC, Laara E, Koivuranta M, Greim CA, Roewer N. A simplified risk score for predicting postoperative nausea and vomiting: conclusions from cross-validations between two centers. Anesthesiology. 1999 Sep;91(3):693-700. doi: 10.1097/00000542-199909000-00022. PMID 10485781
- [Result] Kim SH, Oh YJ, Park BW, Sim J, Choi YS. Effects of single-dose dexmedetomidine on the quality of recovery after modified radical mastectomy: a randomised controlled trial. Minerva Anestesiol. 2013 Nov;79(11):1248-58. Epub 2013 May 23. PMID 23698545